CLINICAL TRIAL: NCT05246670
Title: Treatment of Established Chemotherapy-Induced Neuropathy With N-Palmitoylethanolamide, a Cannabimimetic Nutraceutical: A Randomized Double-Blind Phase II Pilot Trial
Brief Title: PEA for the Relief of Chemotherapy-Induced Peripheral Neuropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ACCRU-SC-2102; NCI-2022-00002 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-SC-2102 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2022-02-11; First posted 2022-02-18 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — palmidrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BID placebo (Placebo Comparator): Patients receive placebo PO BID for 8 weeks.
  Interventions: Drug: Placebo Administration; Other: Quality-of-Life Assessment
- Higher-dose PEA (Experimental): Patients receive PEA PO BID for 8 weeks as long as there is not any unacceptable toxicity.
  Interventions: Drug: Palmidrol; Other: Quality-of-Life Assessment
- Lower-dose PEA (Experimental): Patients receive PEA PO QD for 8 weeks as long as there is not any unacceptable toxicity.
  Interventions: Drug: Palmidrol; Other: Quality-of-Life Assessment
- QD placebo (Placebo Comparator): Patients receive placebo PO QD for 8 weeks.
  Interventions: Drug: Placebo Administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Palmidrol — Given PEA PO
  Other Names: N-Palmitoyl Ethanolamide; N-Palmitoylethanolamide; OptiPEA; Palmitoyl Ethanolamide; Palmitoylethanolamide; PEA
  Arms: Higher-dose PEA; Lower-dose PEA
Drug: Placebo Administration — Given PO
  Arms: BID placebo; QD placebo
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial tests whether PEA works to relieve the symptoms of chemotherapy-induced peripheral neuropathy in patients with cancer. Chemotherapy-induced peripheral neuropathy refers to a nerve problem that causes pain, numbness, tingling, or muscle weakness in different parts of the body, and is caused by chemotherapy. PEA may be useful against bothersome nerve symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To look for evidence of the efficacy of PEA (N-palmitoylethanolamide) at two different doses relative to placebo responses, as a treatment for chemotherapy-induced neuropathy (CIPN).

SECONDARY OBJECTIVES:

I. To assess the safety of PEA at the two study doses. II. To evaluate changes in patient-reported quality of life from baseline to the end of 8 weeks.

EXPLORATORY OBJECTIVES:

I. To explore whether PEA appears to affect cognition in the study patients. II. To explore the weekly trajectory of CIPN from baseline to 8 weeks. III. To explore the weekly trajectory of pain using the single-item numerical rating scale from baseline to 8 weeks.

IV. To explore the weekly patient global impression of change in each treatment arm from baseline to 8 weeks.

V. To explore the weekly chemotherapy induced peripheral neuropathy in each treatment arm from baseline to 8 weeks.

VI. To explore the PEA effects on CIPN20 between two PEA dosage arms. VII. To explore the number of recurrent cancer events by study arm. VIII. To explore the overall survival by study arm.

OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I: Patients receive PEA orally (PO) once daily (QD) for 8 weeks as long as there is not any unacceptable toxicity.

ARM II: Patients receive PEA PO twice daily (BID) for 8 weeks as long as there is not any unacceptable toxicity.

ARM III: Patients receive placebo PO QD for 8 weeks.

ARM IV: Patients receive placebo PO BID for 8 weeks.

After completion of study intervention, patients are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2

  * NOTE: Patients with a history of metastatic cancer or an ECOG performance status of 2 must have laboratory (lab) work completed =< 28 days prior to registration
* Pain, numbness, tingling or other symptoms of CIPN of >= 3 months (90 days) duration for which the patient is seeking an intervention
* Neurotoxic chemotherapy must have been completed >= 3 months (90 days) prior to registration and there must be no further planned neurotoxic -chemotherapy for > 2 months after registration Note: The study is limited to those with taxane- and/or platinum-based neuropathy
* Patient must note tingling, numbness or pain symptoms of at least a four out of ten =< 7 days prior to registration.

  * Note: On a 0-10 scale where zero was 'no problem' and ten being 'as bad a problem that could be imagined': how much of a problem has numbness, tingling, and/or pain in your fingers and/or toes been in the past week?
* Patient must be able to speak, read and comprehend English
* For women of childbearing potential only, a negative urine or serum pregnancy test done =< 14 days prior to registration is required

  * A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

    * NOTE: If the urine test cannot be confirmed as negative, a serum pregnancy test will be required
* Life expectancy >= 6 months
* Platelet count > 100,000/mm^3

  * NOTE: Patients with a history of metastatic breast cancer or an ECOG performance status of 2 must have this lab completed =< 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1,000/mm^3

  * NOTE: Patients with a history of metastatic breast cancer or an ECOG performance status of 2 must have this lab completed =< 28 days prior to registration
* Hemoglobin > 11 g/dL

  * NOTE: Patients with a history of metastatic breast cancer or an ECOG performance status of 2 must have this lab completed =< 28 days prior to registration
* Serum transaminase (alanine aminotransferase [ALT] or aspartate aminotransferase [AST]) =< 1.2 x upper limit of normal (ULN)

  * NOTE: Patients with a history of metastatic breast cancer or an ECOG performance status of 2 must have these labs completed =< 28 days prior to registration
* Alkaline phosphatase =< 1.2 x ULN

  * NOTE: Patients with a history of metastatic breast cancer or an ECOG performance status of 2 must have this lab completed =< 28 days prior to registration
* Serum creatinine =< 1.2 x ULN

  * NOTE: Patients with a history of metastatic cancer or an ECOG performance status of 2 must have this lab completed =< 28 days prior to registration
* Able to swallow oral medication
* Provide written informed consent =< 28 days prior to registration

Exclusion Criteria:

* Currently receiving neurotoxic chemotherapy for a second cancer or recurrence of the primary cancer
* Impaired decision-making capacity (such as with a diagnosis of dementia or memory loss)
* Evidence of residual cancer, per routine clinical practice-based parameters
* Comorbid conditions:

  * Previous diagnosis of diabetic or another non chemotherapy induced peripheral neuropathy
  * Previous history of peripheral neuropathy prior to receiving neurotoxic chemotherapy
  * Neuropathy from human immunodeficiency virus (HIV) infection. Note: Patients with HIV infections are eligible as long as they do not have a neuropathy from their viral illness
* Concurrent use of a cannabis product (tetrahydrocannabinol [THC] and/or cannabidiol [CBD]). Patients should have discontinued these products >= 4 weeks prior to registration
* Current or previous use of PEA
* Currently receiving or planning to start any of the following agents: opioids, duloxetine, gabapentin or pregabalin. Patients are eligible if they discontinue these medications >= 1 week prior to registration
* Any of the following because the study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2026-02-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mellar P Davis, Principal Investigator — Academic and Community Cancer Research United
Locations (10):
- United States (10):
  - Middlesex Hospital, Middletown, Connecticut
  - Carle Cancer Center NCI Community Oncology Research Program, Urbana, Illinois
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Geisinger Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Lower-dose PEA: Patients receive PEA PO QD for 8 weeks as long as there is not any unacceptable toxicity.> > Palmidrol: Given PEA PO>
  > Quality-of-Life Assessment: Ancillary studies
- Higher-dose PEA: Patients receive PEA PO BID for 8 weeks as long as there is not any unacceptable toxicity.> > Palmidrol: Given PEA PO>
  > Quality-of-Life Assessment: Ancillary studies
- QD Placebo: Patients receive placebo PO QD for 8 weeks.> > Placebo Administration: Given PO>
  > Quality-of-Life Assessment: Ancillary studies
- BID Placebo: Patients receive placebo PO BID for 8 weeks.> > Placebo Administration: Given PO>
  > Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Lower-dose PEA | Higher-dose PEA | QD Placebo | BID Placebo
Started | 29 | 30 | 14 | 15
Completed | 25 | 27 | 13 | 14
Not Completed | 4 | 3 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lower-dose PEA | Higher-dose PEA | QD Placebo | BID Placebo | Total
Number analyzed (Participants) | 29 | 30 | 14 | 15 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (7.96) | 60 (10.11) | 56.9 (8.47) | 67.3 (6.05) | 62.7 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 11 | 12 | 71
  Male | 5 | 6 | 3 | 3 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 27 | 27 | 12 | 15 | 81
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 1 | 2 | 13
  White | 22 | 25 | 12 | 13 | 72
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 14 | 15 | 88
Prior Chemotherapy [Count of Participants; unit: Participants]
  Any Taxane +/- carboplatin +/- other agents | 21 | 21 | 10 | 11 | 63
  Oxaliplatin based | 8 | 8 | 4 | 4 | 24
  Other (never received a taxane nor oxaliplatin) | 0 | 1 | 0 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (8.62) | 31.3 (6.81) | 35.1 (8.74) | 31.0 (7.78) | 32.1 (7.90)
ECOG Performance Status [Count of Participants; unit: Participants] — 0 - Fully active, able to carry on all pre-disease performance without restriction; 1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours; 3 - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair; 5 - Dead
  Participants
    0 | 14 | 14 | 8 | 7 | 43
    1+ | 15 | 16 | 6 | 8 | 45

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Quality of Life Questionnaire - Chemotherapy-Induced Peripheral Neuropathy 20 (CIPN20) Score
Description: Will be scored and summarized at each time point for each patient. The change from baseline to 8 weeks will then be calculated for each patient. The mean, standard deviation, and median (range) of the change will be calculated for each PEA arm and the combined placebo arm. The difference in change scores between each PEA arm and the combined placebo will be estimated along with a 95% confidence interval. For the primary analysis, the CIPN20 analysis dataset will include all eligible patients who are randomized, initiated treatment, and completed the baseline questionnaire. For patients who go off protocol treatment before 8 weeks, the score at their final observation will be used to calculate the change. The CIPN20 includes 20 items, each asking a participant to rate their experience with certain symptoms from 1 to 4, with 1 being no difficulty with the symptom and 4 being the most difficulty with the symptom. Answers are then summed to give a total score from 20 to 80.
Time Frame: 8 weeks
Population: All evaluable participants were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lower-dose PEA: Patients receive PEA PO QD for 8 weeks as long as there is not any unacceptable toxicity.
  >
  > Palmidrol: Given PEA PO
  >
  > Quality-of-Life Assessment: Ancillary studies
- Higher-dose PEA: Patients receive PEA PO BID for 8 weeks as long as there is not any unacceptable toxicity.
  >
  > Palmidrol: Given PEA PO
  >
  > Quality-of-Life Assessment: Ancillary studies
- Combined Placebo: Patients receive placebo PO QD or BID for 8 weeks. >
  > Placebo Administration: Given PO
  >
  > Quality-of-Life Assessment: Ancillary studies
Arm/Group | Lower-dose PEA | Higher-dose PEA | Combined Placebo
Number analyzed (Participants) | 27 | 30 | 28
units on a scale | -4.2 (5.42) | -6.3 (12.24) | -6.4 (7.50)
Statistical Analysis 1: Comparison: Lower-dose PEA vs Combined Placebo; Test type: Superiority; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [-1.33 to 5.74]
Statistical Analysis 2: Comparison: Higher-dose PEA vs Combined Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-5.23 to 5.41]
Statistical Analysis 3: Comparison: Lower-dose PEA vs Higher-dose PEA; Test type: Superiority; Mean Difference (Final Values) = 2.11, 95% CI 2-sided [-2.87 to 7.09]

2. Secondary Outcome: Number of Participants Experiencing Grade 3+ Adverse Events
Description: Adverse events by patient will be summarized by frequencies and severity using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. The proportion of patients who experience at least one grade 3+ adverse event (regardless of attribution) will be reported. The overall adverse event rates for grade 3 or higher adverse events will be compared across the three arms (the two PEA arms and combined placebo).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Combined Placebo: Patients receive placebo PO QD or BID for 8 weeks.> > Placebo Administration: Given PO>
  > Quality-of-Life Assessment: Ancillary studies
Arm/Group | Lower-dose PEA | Higher-dose PEA | Combined Placebo
Number analyzed (Participants) | 29 | 30 | 29
Participants | 2 | 0 | 2

3. Secondary Outcome: Mean Change of Quality of Life
Description: Will be assessed by Question 3, patient-reported outcomes-quality of life (PRO-QOL). The mean and standard deviation of the change will be reported for each PEA arm and the combined placebo arm. Additional analysis using data collected from the Symptom Experience Diary may be performed. For patients who go off protocol treatment before 8 weeks, the question 3 response at their final observation will be used to calculate the change. For patients who do not have any post baseline data, they will be considered to have no change from baseline. Question 3 of the PRO-QOL is a 10 point scale asking participants to rate their quality of life, with 0 being the worst and 10 being the best.
Time Frame: 8 weeks
Population: All evaluable participants were included in analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lower-dose PEA | Higher-dose PEA | Combined Placebo
Number analyzed (Participants) | 27 | 30 | 28
units on a scale | 0.6 (2.71) | 0.6 (2.73) | -0.6 (1.91)

4. Other Pre Specified Outcome: Change in the Two Cognitive Items of the Cognitive Functioning Assessment
Description: Will be summarized by mean (SD) and median (range) by treatment arm and the combined placebo arm. The difference in change score will be estimated along with the 95% confidence interval.
Time Frame: Baseline up to 8 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Weekly CIPN20 Scores
Description: Will be summarized at each time point by mean (SD) and median (range) and will be plotted longitudinally by treatment arm and the combine placebo arm.
Time Frame: Baseline up to 8 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Weekly Pain Scores
Description: as for outcome 5
Time Frame: Baseline up to 8 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Items of the Global Impression of Change Tool
Description: Will be summarized by frequency (percentage) of each level at each time point for each treatment arm and the combine placebo arm. Bar plots for each PEA arm and the combined placebo arm of frequency over time will be> constructed.
Time Frame: Baseline up to 8 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Chemotherapy Induced Peripheral Neuropathy Assessment Tool
Description: Will be summarized by mean (SD) and median (range) at each time point for each treatment arm and the combine placebo arm.
Time Frame: Baseline up to 8 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: CIPN20 Score
Description: Will be calculated for each patient. The mean and standard deviation of the change will be calculated for each PEA arm. The difference in CIPN20 change scores between the two PEA dosage arms will be estimated along with a 95% confidence interval.
Time Frame: Baseline up to 8 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Disease Recurrence
Description: The number of events and percentage will be reported by each PEA arm and combined placebo arm. No hypothesis test will be performed between arms.
Time Frame: At 6 and 12 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Overall Survival (OS)
Description: For each PEA arm and combined placebo arm, the distributions of OS time will be estimated using the Kaplan-Meier method. Log-rank test will be used to compare the survival distributions between each PEA and the combined placebo arm.
Time Frame: From registration to death due to any cause, assessed up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Lower-dose PEA | Higher-dose PEA | QD Placebo | BID Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/29 | 0/30 | 2/14 | 0/15
Other Adverse Events (participants affected / at risk) | 8/29 | 6/30 | 3/14 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower-dose PEA (N=29) | Higher-dose PEA (N=30) | QD Placebo (N=14) | BID Placebo (N=15)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower-dose PEA (N=29) | Higher-dose PEA (N=30) | QD Placebo (N=14) | BID Placebo (N=15)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (3) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT05246670/Prot_SAP_000.pdf